CLINICAL TRIAL: NCT03670888
Title: "A Multicenter, Randomized, Double-blind, Parallel-controlled Trial to Compare the Bioequivalence and Safety of the Recombinant Human-Mouse Chimeric Anti-CD20 Monoclonal Antibody Injection (JHL1101) and Rituximab Injection in CD20 Positive B Cell Lymphoma Patients"
Brief Title: A Study to Compare the Bioequivalence and Safety of JHL1101 and Rituximab in CD20 Positive B Cell Lymphoma Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The development was stopped due to company's strategy consideration
Sponsor: JHL Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JHL-CLIN-1101-02
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- JHL1101 (Experimental): Single dose IV infusion of 375 mg/m2 of JHL1101
  Interventions: Biological: JHL1101
- Rituxan (Active Comparator): Single dose IV infusion of 375 mg/m2 of Rituximab
  Interventions: Biological: Rituximab

INTERVENTIONS:
Biological: JHL1101 — 100 mg/10 mL solution in a single-use vial
  Arms: JHL1101
Biological: Rituximab — 100 mg/10 mL solution in a single-use vial
  Arms: Rituxan

SUMMARY:
This is a multicenter, randomized, double-blind, parallel group study to compare the PK, safety, tolerability, immunogenicity and PD of JHL1101 vs Rituxan in subjects with CD20-positive B cell lymphoma. The study duration is 13 weeks. Approximately 128 eligible subjects will be randomized in a 1:1 ratio to receive either JHL1101 (n=64) or Rituxan (n=64). Each subject will receive one intravenous (IV) infusions of the investigational product (IP) at the dose of 375mg/m2 on Day 1. Assessments of PK, safety, tolerability, immunogenicity, PD, and efficacy will be collected over the following 13-week period.

ELIGIBILITY:
Inclusion Criteria:

1. CD20-positive B-cell lymphoma.
2. Obtained CR (complete remission) or CRu (uncertain complete remission) after the prior therapy
3. 18 years to 75 years
4. Signed an informed consent
5. Adequate organ function, including the following

   * Absolute neutrophil count (ANC) ≥ 1,500/uL; platelet count ≥ 75,000/uL; hemoglobin ≥ 8 g/dL
   * Total bilirubin ≤ 1.5 times the upper limit of normal (ULN), aspartate transaminase (AST) and/or alanine aminotransferase (ALT) ≤ 2.5 times ULN
   * Serum creatinine ≤ 1.5 times the ULN
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
7. Chemotherapy: must not have received within 8 weeks of entry onto this study
8. Radiotherapy: must not have received within 4 weeks of entry onto this study
9. Recovery (to baseline or to Grade 1 or less) from prior treatment-related toxicities except alopecia
10. Aagreement to practice contraception
11. More than 6 months life expectancy.

Exclusion Criteria:

1. Received any investigational drug within 28 days prior to study enrollment
2. Received blood transfusion or any therapies with erythropoietin (EPO), granulocyte-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF) within 14 days prior to study enrollment
3. Received previous immunotherapy
4. Received or plan to receive a live vaccine within 28 days of study enrollment
5. Major surgery within 28 days of study enrollment
6. Received systemic steroid therapy with 28 days of study enrollment
7. Received or plan to receive the hematopoietic cell transplant
8. History of gastrointestinal perforation and/or fistula within 6 months prior to study enrollment
9. Known allergic reactions against monoclonal antibody or rituximab.
10. Received rituximab or other anti-CD20 monoclonal antibody
11. Blood concentration of rituximab > 10 ug/mL during screen visit
12. Human immunodeficiency virus (HIV) positive
13. Hepatitis C virus (HCV) antigen and antibody positive
14. Hepatitis B virus surface antigen (HBsAg) positive
15. Body Mass Index (MBI) ≥ 28 kg/m2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

PRIMARY OUTCOMES:
AUC0~t | 91 days
  Area under the concentration-time curve (AUC) from time 0 (predose) of the first infusion on Day 1 to the last quantifiable concentration

SECONDARY OUTCOMES:
AUC0-∞ | 91 days
  AUC from time 0 of the first infusion on Day 1 extrapolated to infinity
Cmax | 91 days
  Maximum concentration after infusion

CONTACTS AND LOCATIONS:
Overall Officials: Lu-Gui Qiu, MD, Principal Investigator — Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (2):
- China (2):
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No